CLINICAL TRIAL: NCT05367128
Title: Effects of Dual Task Prioritization Training on Dual Task Walking in Older People: A Single-blinded Randomized Controlled Trial
Brief Title: Effects of Dual Task Prioritization Training on Dual Task Walking in Older People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Ray-Yau Wang, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YM111015F
Record Dates: First submitted 2022-04-12; First posted 2022-05-10 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Healthy; Older People
Keywords: Older people; Prioritization strategy; Dual task walking; Dual task walking performance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Posture-focus group (Experimental): Participants will be instructed to pay most attention to practice the posture task during training
  Interventions: Other: Dual task training
- Supraposture-focus group (Experimental): Participants will be instructed to pay most attention to practice the cognitive task during training
  Interventions: Other: Dual task training
- Control group (Active Comparator): Participants will not be receive any instruction to prioritize either task
  Interventions: Other: Dual task training

INTERVENTIONS:
Other: Dual task training — All participants will receive cognitive dual task training for 30 min/session, 2-3 sessions/week for 4-6 weeks (a total of 12 sessions). The cognitive dual task training includes 15 min of cognitive task combining with standing task and 15 min of cognitive task combining with walking task. The differences among group are the instructions of task prioritization given by the therapist

SUMMARY:
The purpose of this single-blinded three-armed randomized controlled trial is to investigate the effect of different task prioritization during dual task training on dual task performance.

DETAILED DESCRIPTION:
Introduction: Many activities of daily livings involve performing two tasks simultaneously, i.e. dual tasking. Performing dual task increases the demand on attentional resources, which may further decrease the dual task performance, especially in older adults. According to capacity sharing theory, the two tasks compete and influence with each other due to limited attention and information processing capacity. It has been noted that task prioritization during dual tasking may influence the dual task performance. Previous study indicated that supraposture-focus strategy resulted in better posture and task performance in older people. On the other hand, it is known that dual task training improved dual task performance. However, the effects of applying task prioritization during dual task training have not yet been investigated. Therefore, the purpose of this study is to investigate the effect of different task prioritization during dual task training on dual task performance.

Methods: Participants will be randomized into three groups: posture-focus, supraposture-focus and control group. Participants will receive a total of 12 sessions of cognitive dual task training with different prioritization strategies, i.e. prioritization on posture, cognitive or neither task. Walking and task performance during dual task walking, executive function, and balance performance will be assessed before and after the interventions (pre- and post-test).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years old
* MMSE scores > 24

Exclusion Criteria:

* Unstable health conditions
* Any neurological, psychological disease or diagnosis of learning disability which interferes the participation in this study

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Dual task walking performance assessment- speed (m/s) | Change from baseline dual task walking speed and up to 6 weeks (pre- and post-test)
  Using GaitUp system to evaluate gait speed during cognitive and motor dual task walking
Dual task walking performance assessment- cadence (steps/min) | Change from baseline dual task walking cadence and up to 6 weeks (pre- and post-test)
  Using GaitUp system to evaluate cadence during cognitive and motor dual task walking
Dual task walking performance assessment- stride length variability (CV, %) | Change from baseline dual task walking stride length variability and up to 6 weeks (pre- and post-test)
  Using GaitUp system to evaluate stride length variability during cognitive and motor dual task walking
Dual task walking performance assessment- stride time variability (CV, %) | Change from baseline dual task walking stride time variability and up to 6 weeks (pre- and post-test)
  Using GaitUp system to evaluate stride time variability during cognitive and motor dual task walking
Rate of dual task cost- gait speed (%) | Change from baseline dual task cost and up to 6 weeks (pre- and post-test)
  Using the dual and single task walking speed to calculate the dual task cost of gait speed

SECONDARY OUTCOMES:
Trail Making Test | Change from baseline Trail Making Test and up to 6 weeks (pre- and post-test)
  Use Trail Making Test (TMT)-Chinese version to indicate executive function. The duration for completing the test will be measured, and the shorter duration means the better executive function.
Berg Balance Scale | Change from baseline Berg Balance Scale and up to 6 weeks (pre- and post-test)
  Use Berg Balance Scale (BBS) to assess balance performance. Berg balance scale scoring ranges from 0 to 56. The higher scores indicate better balance performance.
Single task walking performance assessment- speed (m/s) | Change from baseline single task walking speed and up to 6 weeks (pre- and post-test)
  Using GaitUp system to evaluate gait speed during single walking
Single task walking performance assessment- cadence (steps/min) | Change from baseline single task walking cadence and up to 6 weeks (pre- and post-test)
  Using GaitUp system to evaluate cadence during single walking
Single task walking performance assessment- stride length variability (CV, %) | Change from baseline single task walking stride length variability and up to 6 weeks (pre- and post-test)
  Using GaitUp system to evaluate stride length variability during single walking
Single task walking performance assessment- stride time variability (CV, %) | Change from baseline dual task walking stride time variability and up to 6 weeks (pre- and post-test)
  Using GaitUp system to evaluate stride time variability during single walking
Cognitive dual task walking performance assessment- correct number (times) | Change from baseline cognitive dual task walking performance and up to 6 weeks (pre- and post-test)
  The number of the correct answer for serially subtracting "7" from a predefined 3-digit number during cognitive dual task walking task will be recorded.
Motor dual task walking performance assessment- number of go (pieces) | Change from baseline motor dual task walking performance and up to 6 weeks (pre- and post-test)
  The number of successfully transferred go pieces from one side to another during motor dual task walking task will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ray-Yau Wang, PhD, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No